CLINICAL TRIAL: NCT01727752
Title: A Randomized Controlled Trial Comparing Surgical Decompression With an Interlaminar Implant in Patients With Intermittent Neurogenic Claudication Caused by Lumbar Stenosis
Acronym: FELIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paradigm Spine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTR1307
Record Dates: First submitted 2012-11-12; First posted 2012-11-16 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Intermittent Neurogenic Claudication (INC) as a Result of Spinal Stenosis
MeSH Terms: interventions — Decompression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical decompression (Active Comparator): Surgical decompression
  Interventions: Procedure: Decompression
- coflex Interlaminar Technology (Active Comparator): Surgical decompression followed by implantation of coflex Interlaminar Technology.
  Interventions: Procedure: Decompression

INTERVENTIONS:
Procedure: Decompression

SUMMARY:
A Randomized, Blinded Comparison of Surgical Intervention with the Coflex® Interspinous Implant versus Surgical Decompression for Patients with Intermittent Neurogenic Claudication caused by Lumbar Stenosis

DETAILED DESCRIPTION:
In this investigation, it will be investigated whether the effectiveness of surgical intervention with Coflex® is equivalent to surgical decompression after 12 months in people with intermittent claudication. The main advantage of coflex® might be a faster recovery after surgery, but after long term follow-up it is unknown if this treatment effect remains. Therefore in addition, it will be investigated whether surgical intervention with coflex® is more effective than surgical decompression on short-term follow-up (8 weeks to 6 months) and whether surgical intervention with coflex® is more cost-effective after 12 months than surgical decompression.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* is 40 to 85 years old at time of surgery
* has INC, as noted by leg/buttock/groin pain with or without back pain. Leg/buttock/groin pain needs to be strongly relieved when flexed such as when sitting in a chair
* has received at least three months of conservative care therapy which may have included, but is not limited to, physical therapy, bracing, systemic and/or injected medications
* has a regular indication for surgical intervention of INC
* has a narrowed lumbar spinal canal, nerve root canal or intervertebral foramen at one or two levels confirmed by MRI
* is physically and mentally willing and able to comply with, or has a caregiver who is willing and able to comply with, the post-operative evaluations.

Exclusion Criteria:

* has cauda equina syndrome defined as neural compression causing neurogenic bowel (rectal incontinence) or bladder dysfunction (bladder retention or incontinence)
* has Paget's disease, severe osteoporosis or metastasis to the vertebrae
* has significant scoliosis (Cobb angle > 25 degrees)
* has a Body Mass Index (BMI) > 40 kg/m2
* has had any surgery of the lumbar spine
* has degenerative spondylolisthesis > grade 1 (on a scale 1 to 4) at the affected level
* has significant instability of the lumbar spine
* has severe comorbid conditions that will increase the risk to the patient or interfere with the evaluability of this study
* has a fused segment at the indicated level.
* has a herniated disk on the level of interest

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2007-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Zurich Claudication Questionnaire (ZCQ) | 5 years
  ZCQ is a scale that measures physical function, symptom severity, and patient satisfaction for patients with spinal stenosis.

SECONDARY OUTCOMES:
EuroQOL (EQ-5D) | 5 years
  The EuroQol (EQ-5D) will be used for the cost utility analysis at the end of the investigation.
MRDQ | 5 years
  The 23-points MRDQ is the most widely used patient-assessed measure of health outcome for low back pain.
SF-36 | 5 years
  The SF-36 questionnaire relates to the analysis of the general functional status and Quality of Life of patients.
McGill Pain Questionnaire | 5 years
  The McGill questionnaire measures the quality aspect of pain, next to the intensity of pain.
VAS Leg Pain | 5 years
  Improvement of the Visual Analog Scale (VAS) for leg pain (on the 100 mm scale) compared to control group
Re-operations, revisions, and major complications | 5 years
  Assessment of revisions, removals, re-operations, and major device-related complications.
Radiographic Assessment | 12 months
  Radiographic Assessment of coflex and control group

CONTACTS AND LOCATIONS:
Locations (13):
- Netherlands (13):
  - Sint Lucas Andreas Ziekenhuis, Amsterdam
  - Reinier De Graaf Gasthuis, Delft
  - Groene Hart Ziekenhuis, Gouda
  - Medical Center Alkmaar, Holland
  - Diaconessenhuis, Leiden
  - Leiden University Medical Center, Leiden
  - Rijnland ziekenhuis,, Leiderdorp
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Vlietland Ziekenhuis, Schiedam
  - Bronovo Ziekenhuis, The Hague
  - HAGA ziekenhuis, The Hague
  - Medical Center Haaglanden, The Hague/Leidschendam
  - Isala Klinieken, Zwolle